CLINICAL TRIAL: NCT01933113
Title: Effects of Deep Brain Stimulation of the Lateral Hypothalamic Area on Weight Change and Metabolic Rate
Brief Title: Deep Brain Stimulation Effects on Weight Change and Metabolic Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, donald whiting, Principal Investigator, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBS 5583
Record Dates: First submitted 2013-08-23; First posted 2013-09-02 (Estimated); Results first posted 2019-01-08 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: Obesity; Deep Brain Stimulation; LHA
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DBS of the Lateral Hypothalamic Area (Experimental): Single Arm: Deep Brain Stimulation of LHA for maximum RMR On days 1-4, subjects stayed in the inpatient unit to have metabolic weight, temperature, and resting metabolic rate (RMR) measured at different settings.
  Metabolic testing RMR measurement: A clear plastic hood was placed over the head and chest Oxygen intake and carbon dioxide out-put were measured to determine how many calories were burned during the next 15-30 minutes. Each hour for the next seven hours, DBS settings were changed and the above process was repeated. On Day 4, a DXA scan was performed to assess body composition. Primary endpoint is the determination of optimal settings
  Interventions: Device: Deep Brain Stimulation of the Lateral Hypothalamic Area

INTERVENTIONS:
Device: Deep Brain Stimulation of the Lateral Hypothalamic Area — Deep Brain Stimulation of the Lateral Hypothalamic Area
  Other Names: Devices used in this protocol:; Medtronic Activa TM SC model # 37603; Medtronic DBS lead model # 3389; Medtronic Extension model # 37086-60

SUMMARY:
This study focuses on lateral hypothalamic area (LHA) deep brain stimulation (DBS) for severe obesity. In a previous pilot study, three subjects were implanted with a DBS electrode into the LHA under an Investigational Device Exemption (IDE) and IRB approved study at West Virginia University. That study demonstrated the safety of DBS of the LHA in these patients. These patients, who met the enrollment criteria of having prior placement of LHA DBS in accordance with previous study protocol, were eligible for this study with a goal of determining optimal DBS settings.

DETAILED DESCRIPTION:
The goal of this study was to investigate changes in Resting Metabolic Rate (RMR) at different settings during stimulation of the LHA with DBS and to find the optimal setting for increasing the RMR in two patients that previously were implanted. Although 3 subjects had undergone placement of the DBS electrode in the pilot study, one subject was withdrawn from this study due to a lead breakage and medical instability pertaining to an unrelated abdominal infection.

Each subject utilized the metabolic chambers and Deltatrac II Metabolic Carts (SensorMedics Corporation, Anaheim, California or Datex-Ohmeda, Helsinki, Finland) at Pennington Biomedical Research Center (PBRC), in Baton Rouge, Louisiana to objectively measure the correlation of their metabolic rate to various novel settings on the DBS for a one week period.

The schedule for the metabolic testing included: Day 0 baseline overnight chamber with no stimulation. Days 1-4 Resting metabolic rate (RMR) will be performed hourly with variable LHS DBS settings. The settings will be changed approximately every 15 minutes after the DBS settings are changed. Day 4 overnight chamber at ideal metabolic rate setting. After RMR test on Day 4, the subject will have a dual-energy x-ray absorptiometry (DXA) scan performed to assess body composition.

Subjects were also be seen in clinic as often as every month but no less than every 3 months to assess changes in weight until the study ended.

ELIGIBILITY:
Inclusion Criteria:

* Prior placement of LHA DBS in accordance with previous study protocol

Exclusion Criteria:

* Not a participant of the original LHA DBS study
* Prior brain surgery, excluding the placement of LHA DBS
* Taking medications with a recognized adverse event of weight change.
* Diagnosis of a neurological disorder, such as multiple sclerosis or stroke.
* Concurrent use of weight-loss prescription drug therapy or the use of over- the-counter weight loss preparations.
* Unable to participate in scheduled study visits

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald M Whiting, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny Health Network, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Whiting DM, Tomycz ND, Bailes J, de Jonge L, Lecoultre V, Wilent B, Alcindor D, Prostko ER, Cheng BC, Angle C, Cantella D, Whiting BB, Mizes JS, Finnis KW, Ravussin E, Oh MY. Lateral hypothalamic area deep brain stimulation for refractory obesity: a pilot study with preliminary data on safety, body weight, and energy metabolism. J Neurosurg. 2013 Jul;119(1):56-63. doi: 10.3171/2013.2.JNS12903. Epub 2013 Apr 5. PMID 23560573
- [Background] Whiting AC, Sutton EF, Walker CT, Godzik J, Catapano JS, Oh MY, Tomycz ND, Ravussin E, Whiting DM. Deep Brain Stimulation of the Hypothalamus Leads to Increased Metabolic Rate in Refractory Obesity. World Neurosurg. 2019 Jan;121:e867-e874. doi: 10.1016/j.wneu.2018.10.002. Epub 2018 Oct 11. PMID 30315980

RESULTS

PARTICIPANT FLOW:
Groups:
- Single arm: DBS of the LHA
  Deep Brain Stimulation of the Lateral Hypothalamic Area
Period: Overall Study
Arm/Group | Single arm
Started | 3
Completed | 2
Not Completed | 1
Not completed — Fractured nonfunctioning lead. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject was withdrawn due to a lead breakage and medical instability pertaining to an unrelated abdominal infection.
  Participants
    Female | 2
    Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
BMI [Count of Participants; unit: Participants] — Chronic obesity as defined as a BMI over 40 Population: One subject was withdrawn due to lead fracture and unrelated abdominal infection leaving 2 evaluable subjects
  Participants
    number analyzed (Participants) | 2
    (all) | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Metabolic Rate
Description: Metabolic rate of subjects will be measured while at Pennington Biomedical Research Center. Percentage of change in these parameters will be measured.
Time Frame: One week of testing for each subject.
Measure: Median (Standard Deviation); unit: percentage of increase in REM and SEE
Arm/Group | Single arm
Number analyzed (Participants) | 2
percentage of increase in REM and SEE
  Sleep Energy Expenditure (SEE) | 7.6 (3.9598)
  Resting Metabolic Rate (RMR) | 18 (2.8284)

ADVERSE EVENTS:
Time Frame: Subjects were followed for a total of one week
Groups:
- Single arm: Deep Brain Stimulation (DBS) of the Lateral Hypothalamic Area (LHA)
Arm/Group | Single arm
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes